CLINICAL TRIAL: NCT04468763
Title: Cardiac Biomarkers in Preeclampsia: Prediction of Disease and the Risk of Future Cardiovascular Events in Survivors
Acronym: PreeclampBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Babcock University (Other)
Responsible Party: Sponsor
Other Study IDs: BUHREC014/19; OOUTH/HREC/248/2019AP (Other: OOTH Sagamu)
Record Dates: First submitted 2020-01-27; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-01

CONDITIONS: Preeclampsia; Eclampsia
Keywords: Cardiac biomarkers; Prediction; Preeclampsia; Stroke
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After explaining the procedure with the aid of the subject information form, obtaining consent and completing the history segments of the proforma, 10ml of venous blood samples would be obtained from the participants prior to the commencement of any intravenous therapy. This sample would be collected from the contra-lateral upper limb of patients who are already on intravenous infusion. The venous blood would be aspirated from the participant's ante-cubital vein and placed in a lithium heparin vacuum tube (5mls) and a plain anticoagulant-free bottle (5mls). At the time of blood collection, a drop of blood would be made on a filter paper for genetic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SUMMARY Background: Improvements in the management and prevention of obstetric haemorrhage and sepsis, in addition to magnesium sulphate for preeclampsia have led to significant reduction in global maternal mortality rates; thus leaving increasing number of survivors of preeclampsia than previously. Preeclampsia is associated with inflammatory changes that alter vascular integrity - an effect which may persist beyond pregnancy, resulting in atherosclerosis which predisposes to myocardial ischemia, myocardial infarction and stroke.

Aim: To predict preeclampsia early in pregnancy and detect preeclampsia survivors at risk for future cardiovascular disease and events using cardiac and gene markers.

Methods: a cohort study design with recruitment of participants at 3 stages; in the first trimester of pregnancy, second half and the puerperium. Serum levels of fibrinogen, hsCRP, apoA/apoB, triglycerides and other lipids, in addition to genetic studies would be compared between those with preeclampsia and normal pregnancies, delivered mothers would be followed up from puerperium, upto 5 years.

Data Analysis: would be performed using the Statistical Package for Social Sciences (SPSS) software version 21.0. Numerical data would be expressed as mean ± standard deviation (SD). Results from the two groups of women would be compared using the independent T-test, Analysis of Variance (ANOVA) and the chi-square test while the Mantel Haenszel statistics would be used to determine risks. The level of statistical significance would be set at p-value less than 0.05.

Conclusion: Myocardial ischemia, myocardial infarction and stroke are major causes of sudden death because their precursors; atherosclerosis and hypertension are asymptomatic. Under-utilization of routine health care check further increases the risk of sudden death from these conditions. Preeclampsia is a recognized risk factor and screening of survivors would help to detect women at risk for cardiovascular diseases and offer early preventive care.

DETAILED DESCRIPTION:
Preeclampsia is a disease that is strongly linked with the risk of stroke and other cardiovascular disease. This is a condition with greater prevalence in the Low and middle income countries of the world especially sub-Saharan Africa, where the morbidity and mortality is reportedly higher. Larger numbers of survivors are expected with the rising global gains in maternal mortality reduction associated with preeclampsia. These cardiovascular diseases myocardial ischemia, myocardial infarction and stroke are major causes of sudden death because the precursor conditions; atherosclerosis and hypertension are largely asymptomatic. There are established biomarkers for these conditions which can be used as screening tools. The low utilization of routine health care check and the asymptomatic nature of these events increase the risk of sudden premature death from these conditions. The postnatal period offers a good opportunity for screening for these events to detect women at risk and offer early preventive care.

Preeclampsia is essentially a disease of the trophoblast, it has also been shown to be associated with oxidative stress, a phenomenon, which increases the levels of LDL cholesterol peroxidation, leading to its increased uptake by macrophages, resulting in foam cell formation and atherosclerosis. Preeclampsia is also associated with inflammatory changes that alter vascular integrity - an effect which may persist beyond pregnancy, resulting in atherosclerosis which predisposes to myocardial ischemia, myocardial infarction and stroke.

These changes in the vasculature are asymptomatic and unless hypertension is detected early and vasoprotective or antithrombotic treatment commenced, sudden death may occur from stroke or acute myocardial infarction.

Hypertensive heart disease refers to heart conditions that result from the effect of hypertension. The heart in this instance now works under a higher pressure resulting in the hypertrophy of cardiac muscle, thickening of the cardiac arterial vasculature (leading to coronary arterial disease) and increased risk of myocardial ischemia and infarction. The resulting cardiac muscle dysfunction leads to increasing levels of pro-inflammatory cytokines, which can be detected in the blood stream and whose levels may correlate with the presence and severity of the disease condition. Hypertension has similar effects on the cerebral vasculature, where it can cause vessel rupture resulting in life-threatening intracranial haemorrhage. The vessels under the influence of long standing hypertension may undergo hypertrophy leading to thickening of the vessel wall with narrowing of lumen and then cerebral ischemia, infarction and stroke.

There is a significant reduction in the risk of fatal and non-fatal stroke if hypertension is detected early and effectively controlled with antihypertensive drugs. This preventive strategy has been shown to be of more benefit when commenced at a younger age and especially in women of the black race who are at higher risk and would benefit more.

In the general adult population, lipids and cardiac biomarkers have been shown to predict the occurrence of these cardiovascular events. These biomarkers include: High sensitivity C-reactive Protein (hsCRP), Apolipoproteins (LDL, Apo B-100, Apo A1), Lipoprotein a (Lp(a), Oxidized LDL, Lipoprotein-associated phospholipase (A2-LpPLA2), Sphingosine-1-phosphate (Sph-1-P), small dense low density lipoprotein (sdLDL) and Myeloperoxidase (MPO). A recent systematic review on markers for primary cardiovascular events revealed that in terms of correlation with the development of cardiovascular disease; C-reactive protein, fibrinogen, cholesterol, apolipoprotein B, the apolipoprotein A/apolipoprotein B ratio, high density lipoprotein, and vitamin D, were useful in the prediction of cardiovascular disease, while for primary stroke; fibrinogen and serum uric acid were strong markers.

This study therefore aimed to determine the risk of future cardiovascular disease and events in survivors of preeclampsia using these established biomarkers, in conjunction with testing for gene markers.

Participants would include all consecutive participants who meet the inclusion criteria for each group of study within the 12-month period at all sites. They would be educated about the study and informed consent obtained from them or from relatives (when patient is unable to do so). A 10ml sample of venous blood and a dry blood spot on filter paper would be obtained (by doctors from all the participating sites) from all the participants for assay of cardiac, lipid and gene markers of cardiovascular disease.

At the start of the study, training sessions on the study protocol and monitoring would be held for all team members from the study sites and this would be done fortnightly until completion of study to ensure uniformity.

Blood samples obtained would be centrifuged to obtain plasma and serum at each study site which would then be transported in ice packs department of medical laboratory science of the Babcock University, Ilishan-Remo for assay of lipid and cardiac biomarkers while the genetic studies (DNA extraction and sequencing) would be done at the Centre for Advanced Medical Research and Biotechnology (CAMRAB), laboratory at Babcock University Teaching Hospital, Ilishan-Remo. All samples obtained would be coded such that the laboratory scientist is blinded from the identity of the participants. The results obtained would then be transferred into the pre-labelled proforma where other details of each participant including the biodata and pregnancy history have already been entered. The participants details entered into the proforma would also be entered directly into tablets linked with Redcap mobile application for web hosting, which would then be exported later to SPSS for analysis. Twenty four-hour telephone contact would be maintained with team members from all the study sites involved in the study, through direct phone call and text message. A whatsapp chat group would be created to link all four study sites for easy transmission of information. Twenty four-hour telephone contact would be maintained with team members from all the study sites involved in the study.

The blood samples would be collected into lithium heparin and plain anticoagulant-free containers and transported immediately in an ice container to the laboratory for analysis where they would be centrifuged at 2,500 rpm for 5 minutes, at all sites, before transport of both well labelled supernatant sera in plain bottles and plasma in lithium heparin bottles after decanting from the packed red cells to Babcock University. Serum and plasma aliquots would then be stored at -20ºC in Babcock University until further analysis. The drop of blood spot obtained from each participant would be allowed to air-dry and then safely stored in a cool dry storage refrigerator before transport to CAMRAB, where it would be maintained at -80˚C until gene analysis. Serum and plasma samples that are not used would be stored at -80˚C for 5 years.

Blood pressure measurements would be obtained by a trained nurse at each site with manually operated mercury powered sphygmomanometer and these readings would be taken in the sitting position. The Korotkoff sound V would be taken as the level for diastolic blood pressure in all cases. The blood pressure would then be immediately entered into the study proforma for each participant.

After explaining the procedure with the aid of the subject information form, obtaining consent and completing the history segments of the proforma, 10ml of venous blood samples would be obtained from the participants prior to the commencement of any intravenous therapy. This sample would be collected from the contra-lateral upper limb of patients who are already on intravenous infusion. The venous blood would be aspirated from the participant's ante-cubital vein and placed in a lithium heparin vacuum tube (5mls) and a plain anticoagulant-free bottle (5mls). At the time of blood collection, a drop of blood would be made on a filter paper for genetic analysis.

All participants would be followed up till end of puerperium thus; observation for the development of preeclampsia in women admitted within the first half of pregnancy, those admitted with preeclampsia in pregnancy would be observed for the correlation of preeclampsia severity with the levels of biomarkers and those recruited postpartum would have their levels of cardiac and gene markers compared with those of women who had normal pregnancies. Telephone contact of the participants and their next of kin would be obtained and they or next of kin would be contacted at 1, 2, 5 and 10 year intervals for development of cardiovascular events and repeat serum levels of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women at gestational age less than 20 weeks
* Women with diagnosis of preeclampsia at gestational age 20-41 weeks
* Healthy pregnant women without preeclampsia at gestational age 20-41 weeks
* Women less than one year postpartum with history of preeclampsia or eclampsia in index pregnancy
* Healthy women less than 1 year postpartum with no previous history of preeclampsia or eclampsia

Exclusion Criteria:

* History of chronic hypertension or hypertension before pregnancy
* Patients with cardiac disease
* Patients with renal disease
* Patients with diabetes mellitus
* Patients with connective tissue disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 18-45 years, pregnant after 20 weeks gestational age, or within puerperium, with or treated for preeclampsia or eclampsia.
Study Population: The participants would include 3 groups of women all aged between 18-45 years, recruited from the study sites who give a written informed consent.
  1. Group 1: Pregnant women within the first 20 weeks of gestation who come to register for antenatal care.
  2. Group 2: Pregnant women diagnosed with preeclampsia or eclampsia whose pregnancies are between 20 and 41 weeks.
  3. Group 3: Delivered mothers who are within 1 year post-delivery.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Serum levels of cardiac biomarkers | Baseline
  Serum concentrations of hsCRP, fibrinogen, apoB, lipid profile in mg/dL

SECONDARY OUTCOMES:
Development of cardiovascular events | Year 1, Year 2 and Year 5
  Incidence of hypertension (blood pressure >/=140/90 mmHg), Incidence of stroke (clinical, CT or MRI) and Incidence of myocardial infarction (clinical or ECG) in participants with elevated biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Oladapo Walker, MBBS,PhD, Study Chair — Babcock University
Locations (1):
- Babcock University Teaching Hospital, Sagamu, Ogun State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT04468763/ICF_000.pdf